CLINICAL TRIAL: NCT05993234
Title: A Prospective Non-interventional Study (NIS) of Trastuzumab DeRuxtecan (T-DXd) for Adult Patients With Advanced HER2-pOsitive GaStric or GastroesoPhageal Junction (GEJ) AdEnocarcinoma Who Have Received a PrIor Trastuzumab-based Regimen, Accompanied by a Disease RegistrY of Patients Treated With Conventional Therapies in a Real-world Setting in Europe (PROSPERITY)
Brief Title: A Study of Trastuzumab DeRuxtecan for Patients With Advanced HER2-pOsitive GaStric or GastroesoPhageal Junction AdEnocarcinoma Who Have Received a PrIor Trastuzumab-based Regimen Accompanied by a Disease RegistrY of Patients Treated With Conventional Therapies (PROSPERITY)
Status: Recruiting | Type: Observational
Sponsor: Daiichi Sankyo Europe, GmbH, a Daiichi Sankyo Company (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Other Study IDs: DS8201-0007-NIS-MA
Record Dates: First submitted 2023-08-02; First posted 2023-08-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: HER2-positive Advanced Gastric Cancer; HER2-positive Gastroesophageal Junction Adenocarcinoma
Keywords: HER2-positive Advanced Gastric Cancer; HER2-positive Gastroesophageal Junction Adenocarcinoma; Trastuzumab Deruxtecan; Conventional therapy; ENHERTU®
MeSH Terms: interventions — trastuzumab deruxtecan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trastuzumab deruxtecan (T-DXd): Participants with HER2-positive gastric or gastroesophageal junction adenocarcinoma who will be treated with trastuzumab deruxtecan and part of the enrolled participants will receive conventional therapy. The participants on conventional therapy will be analyzed for exploratory purposes only.
  Interventions: Drug: Trastuzumab deruxtecan

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — This is a non-interventional study and medication will be administered according to the SmPC as local standard of care and as part of the routine clinical practice.
  T-DXd to be administered according to the SmPC. Conventional therapy (eg. platinum-fluoropyrimidine doublet chemotherapy, nivolumab, ramucirumab-paclitaxel, ramucirumab monotherapy, taxane or irinotecan, and pembrolizumab monotherapy) to be administered according to the SmPC.
  Other Names: T-DXd; ENHERTU®

SUMMARY:
Trastuzumab deruxtecan (T-DXD) as monotherapy is indicated for the treatment of adult patients with advanced HER2-positive advanced gastric or gastroesophageal junction (GEJ) adenocarcinoma who have received a prior trastuzumab-based regimen.

This study will assess the effectiveness of T-DXd, patient demographic and clinical characteristics, and treatment patterns in patients with advanced HER2-positive advanced gastric or GEJ adenocarcinoma.

DETAILED DESCRIPTION:
This non-interventional study will investigate the effectiveness of T-DXd, the patients demographic and clinical characteristics, treatment patterns including prophylactic medications and interventions for reduction of serious adverse events (SAEs), serious adverse drug reactions (ADRs) and safety event of interest (SEIs), tolerability, and patient survey of T-DXd, in cases with advanced HER2-positive gastric or GEJ adenocarcinoma receiving T-DXd as second line of treatment and beyond treatment option. Patients will be treated according to the proposed indication statement in the Summary of Product Characteristics (SmPC). No investigational drug will be administered in this study.

Data on conventional therapy (including platinum-fluoropyrimidine doublet chemotherapy, nivolumab, ramucirumab-paclitaxel, ramucirumab monotherapy, taxane or irinotecan, and pembrolizumab monotherapy) will also be collected in a disease registry part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult patient (age ≥ 18 years) with HER2 + advanced gastric or GEJ adenocarcinoma who have received a prior trastuzumab based regimen
* Histological or cytological confirmed diagnosis of advanced HER2 positive gastric cancer or GEJ
* Documented HER2 + status (archival sample or recent sample prior 2L therapy)
* Decision to newly initiate monotherapy T-DXd or conventional therapies per SMPC according to the physician's choice
* Written dated and signed Informed Consent (ICF) to participate in the study

Exclusion Criteria:

* Patients who at time of data collection for this study are participating in or have participated in an interventional study that remains blinded
* Pregnancy or breastfeeding

No specific exclusion criteria are defined, as patients will be treated according to the proposed indication statements in the SmPC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with advanced HER2-positive gastric or GEJ adenocarcinoma who have received a prior trastuzumab-based regimen in a real-world setting in Europe.
Sampling Method: Non-Probability Sample
Enrollment: 257 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Real-World Time to Next Treatment (rwTTNT1) in Participants With HER2-positive Gastric or Gastroesophageal Junction Adenocarcinoma | Baseline up to approximately 2 years

SECONDARY OUTCOMES:
Number of Physician Visits and Treatment Changes in Participants With HER2-positive Gastric or Gastroesophageal Junction Adenocarcinoma | Baseline up to approximately 2 years
Number of Physician-reported Safety Events of Interest in Participants With HER2-positive Gastric or Gastroesophageal Junction Adenocarcinoma (T-DXd only) | Baseline up to approximately 2 years
Number of Participants Receiving Prophylactic and Reactive Treatment Management for Physician-reported Safety Events of Interest in Participants With HER2-positive Gastric or Gastroesophageal Junction Adenocarcinoma (T-DXd only) | Baseline up to approximately 2 years
Real-World Time to Permanent Treatment Discontinuation (rwTTD1) in Participants With HER2-positive Gastric or Gastroesophageal Junction Adenocarcinoma | Baseline up to approximately 2 years
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) Scores in Participants With HER2-positive Gastric or Gastroesophageal Junction Adenocarcinoma | Baseline up to approximately 2 years
  The EORTC QLQ-C30 questionnaire is a cancer-specific quality of life instrument applicable to a broad range of cancer patients. The EORTC QLQ-C30 scales and single-item scales range in score from 0 to 100. A higher score for the functioning scales and global health status denotes a better level of functioning (i.e. a better state of the patient), while higher scores on the symptom and single-item scales indicate a higher level of symptoms (i.e. a worse state of the patient).
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Stomach (EORTC QLQ-STO22) Score in Participants With HER2-positive Gastric or Gastroesophageal Junction Adenocarcinoma | Baseline up to approximately 2 years
  The EORTC QLQ-STO22 is a gastric cancer-specific module which has been developed to measure the quality of life in patients with gastric cancer. The gastric cancer specific questions on the EORTC QLQ-STO22 include four single-item subscales (dry mouth, body image, hair loss and problems with taste) and five multi-item subscales (dysphagia, dietary restriction, pain, upper gastroesophageal symptoms and emotional problems). The EORTC QLQ single-item and multi-item scales range in score from 0 to 100. A higher score on the symptom and single-item scales indicate a higher level of symptoms (i.e. a worse state of the patient)

CONTACTS AND LOCATIONS:
Overall Officials: Global Team Leader, Study Director — Daiichi Sankyo Europe, GmbH, a Daiichi Sankyo Company
Locations (76):
- Austria (9):
  - KABEG Klinikum Klagenfurt am Wörthersee - Landeskrankenanstalten LKH, Klagenfurt
  - Ordensklinikum Linz GmbH Barmherzige Schwestern, Linz
  - Universitätsklinikum St. Pölten - Lilienfeld, Sankt Pölten
  - Medizinische Universität Wien, Vienna
  - St. Josef Krankenhaus GmbH Ein Unternehmen der Vinzenz Gruppe, Vienna
  - Klinik Ottakring, Wilhelminenspital der Stadt Wien, Vienna
  - Kepler Universitätsklinikum, Wels
  - Landesklinikum Wiener Neustadt, Wiener Neustadt
  - Krankenhaus St. Vinzenz in Zams, Zams
- Belgium (11):
  - OLV Hospital Aalst, Aalst
  - Imelda vzw, Bonheiden
  - HUB institut Jules Bordet, Brussels
  - Grand hôpital de Charleroi, Charleroi
  - Antwerp University Hospital, Edegem
  - UZ Gent, Ghent
  - CHU Helora Hospital de La Louvière - Site Jolimont, Haine-Saint-Paul
  - JESSA Hasselt, Hasselt
  - UZ Brussel, Jette
  - UZ Leuven, Leuven
  - AZ Delta, Roeselare
- Germany (25):
  - MVZ am Klinikum Aschaffenburg, Aschaffenburg
  - Universitätsklinikum Augsburg, Augsburg
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Charite Campus Benjamin Franklin, Berlin
  - Klinikum Chemnitz gGmbH, Chemnitz
  - MV-Zentrum für Hämatologie & Onkologie, Cologne
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - University Hospital Essen, Essen
  - Universitaetsklinikum Giessen und Marburg, Standort Giessen, Giessen
  - Alb Fils Kliniken GmbH, Göppingen
  - Hämatologisch-Onkologische Praxis Eppendorf (HOPE), Hamburg
  - Studienzentrum am Raschplatz GbR, Hanover
  - KRH Klinikum Siloah, Hanover
  - Gemeinschaftspraxis Dr. Haytham Kamal / Dr. David C. Dorn, Hanover
  - Städtisches Klinikum Karlsruhe, Karlsruhe
  - ÜBAG MVZ Mitte / MVZ Delitzsch GmbH, Leipzig
  - Praxis Hämatologie und Onkologie Magdeburg, Magdeburg
  - Universitätsklinik für Gastroenterologie, Hepatologie und Infektiologie, Magdeburg
  - Klinikum rechts der Isar der Technischen Universität München, München
  - Pi.Tri-Studien GmbH, Offenburg
  - Klinikum am Steinenberg Reutlingen, Reutlingen
  - Nädler GmbH, Rinteln
  - CaritasKlinikum Saarbrücken, Saarbrücken
  - Praxis Onkologie Rheinsieg, Troisdorf
  - Universitätsklinikum Würzburg (UKW), Würzburg
- Italy (23):
  - AOU delle Marche, Ancona Torrette
  - ASL AT - Presidio Ospedaliero "Cardinal Massaia", Asti
  - IRCCS "S. De Bellis", Castellana Grotte
  - ARNAS Garibaldi - PO Nesima, Catania
  - AOU Careggi, Florence
  - IRCCS AOU San Martino, Genova
  - IRCCS Ospedale San Raffaele, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Azienda Ospedaliero-Universitaria di Modena, Modena
  - A.O.U. Cagliari - Policlinico Universitario Duilio Casula, Monserrato
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Napoli
  - Università degli studi di Napoli Federico II, Napoli
  - Università della Campania 'Luigi Vanvitelli', Napoli
  - AOU Pisana - Stabilimento Santa Chiara, Pisa
  - Azienda Sanitaria Locale di Biella - Ospedale degli Infermi, Ponderano
  - AUSL della Romagna - Ospedale "S. Maria delle Croci" di Ravenna, Ravenna
  - Policlinico Universitario Campus Bio-Medico, Roma
  - AO San Camillo Forlanini, Roma
  - AO San Giovanni Addolorata, Roma
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - AO "Cardinale Giovanni Panico", Tricase
  - ASU FC - Ospedale "Santa Maria della Misericordia", Udine
  - Azienda ULSS 8 Berica - Ospedale San Bortolo, Vicenza
- Portugal (8):
  - ULS Almada-Seixal, Almada
  - USL Braga, Braga
  - ULS Coimbra, Coimbra
  - IPO Lisboa, Lisbon
  - CC Champalimaud, Lisbon
  - Hospital da Luz, Lisbon
  - ULS Santo António, Porto
  - Vila Real, Vila Real

IPD SHARING:
Plan to Share IPD: No